CLINICAL TRIAL: NCT01551160
Title: Impact of a Communication and Team-working Intervention on Performance and Effectiveness of a Medical Emergency Team
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lyell McEwin Hospital (Other Government)
Collaborators: University of Adelaide (Other)
Responsible Party: Principal Investigator, Dr Richard Chalwin, Principal Investigator, Lyell McEwin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RPC1001
Record Dates: First submitted 2012-03-04; First posted 2012-03-12 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Hospital Rapid Response Team
Keywords: Non-technical skills; Crisis resource management; Medical Emergency Team; Rapid Response Team

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medical Emergency Team (Experimental): A communication and team-working initiative
  Interventions: Other: A communication and team-working intervention

INTERVENTIONS:
Other: A communication and team-working intervention — Medical Emergency Team (MET) briefings and formalised handover between MET staff and patient care teams

SUMMARY:
Patients in hospital can have unexpected clinical emergencies. When this occurs the Medical Emergency Team (MET) are called with the intention of resolving the problem. Previous investigations have found that patients who have more than one call during their admission have worse outcomes than patients who only have one call. But it has not been established why.

The aim of this research will be to examine these repeated calls and why patients subject to them go on to have worse outcomes. A predictive model will be developed to identify potential sources of risk. One potential source is poor communication between health care providers. An intervention to improve communication around MET calls may provide benefit to patients and improve outcomes.

DETAILED DESCRIPTION:
This investigation will comprise a mixed methods, before-and-after study. The particulars are:

Format:

1. Before intervention

   1. Analysis of retrospective MET activity and patient outcome data
   2. Surveying of staff for attitudes and perceptions of MET calls
2. Intervention

   1. Twice-daily MET briefing meetings
   2. Formalised handover process for MET calls resulting in patients remaining in their current clinical area
3. After intervention

   1. Analysis of prospective MET activity and patient outcome data
   2. Surveying of staff for attitudes and perceptions of MET calls

Setting:

Lyell McEwin Hospital, a 300 bed, university-affiliated, tertiary, metropolitan hospital located in Adelaide, South Australia. It has comprehensive in-patient medical and surgical services including a Level 3 Intensive Care Unit.

Subjects:

1. Patients - adult in-patients attended by the MET during the study period. This will include patients attended more than once during an admission, as all calls will be a separate datapoint. It is also possible for patients to have more than one admission during the study period, so each admission will be considered discretely.
2. Staff - members of the hospital MET and ward staff that may call the MET. The MET composition is an ICU doctor, ICU nurse, medical registrar, intern and hospital manager. Due to rostering demands, this team is supplied from a pool of staff within each of the representative departments (approximately 10 ICU doctors, 30 ICU nurses, 30 medicine registrars, 36 interns and 8 duty managers).

Data Collection:

1. Characteristics and Outcomes

   1. Per-hospital admission data includes: age, gender, admission diagnosis, admission type, length of stay and mortality
   2. Per-MET call data includes: reason for call, location, duration of call, interventions performed, disposition and mortality
2. Perceptions and Attitudes

   1. Ward staff question including around interactions with MET, involvement during MET calls, experience of repeat calling and reasons for repeat calling
   2. MET questions including around interactions with ward staff, involvement of ward staff during calls and resolution of calls.

ELIGIBILITY:
Inclusions

- Medical Emergency Team (MET) calls

Exclusion Criteria:

* Cancellation of the MET response prior to, or on arrival at, the location of activation
* Calls to patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Multiple Medical Emergency Team calls per patient admission | Measured at time of hospital discharge

SECONDARY OUTCOMES:
Mortality | At time of hospital discharge
Mortality | At completion of Medical Emergency Team call
ICU admission rate | At completion of Medical Emergency Team call
ICU interventions | At completion of Medical Emergency Team call

OTHER OUTCOMES:
Perceptions of Interactions between Medical Emergency Team staff and patient care teams | 1 year
  Both Medical Emergency Team staff and patient care teams will be surveyed separately

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chalwin, FCICM, Principal Investigator — Lyell McEwin Hospital
Locations (1):
- Lyell McEwin Hospital, Elizabeth Vale, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalwin RP, Flabouris A. Utility and assessment of non-technical skills for rapid response systems and medical emergency teams. Intern Med J. 2013 Sep;43(9):962-9. doi: 10.1111/imj.12172. PMID 23611153
- [Derived] Chalwin R, Giles L, Salter A, Kapitola K, Karnon J. Re-designing a rapid response system: effect on staff experiences and perceptions of rapid response team calls. BMC Health Serv Res. 2020 May 29;20(1):480. doi: 10.1186/s12913-020-05260-z. PMID 32471422